CLINICAL TRIAL: NCT02079935
Title: Treatment of Eating Disorders - a Randomised, Controlled, Prospective Study
Brief Title: Treatment of Eating Disorders by Physical Activity and Nutrition Counseling
Acronym: FAKT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: The Norwegian Women´s Public Health Association (Other); University of Tromso (Other)
Responsible Party: Principal Investigator, Professor Jorunn Sundgot-Borgen, Professor, Norwegian School of Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013/344; 2013/1871 (Other Grant/Funding Number: Regional Committees for Medical and Health Research Ethics)
Record Dates: First submitted 2014-02-17; First posted 2014-03-06 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Bulimia Nervosa; Binge Eating Disorder
Keywords: BN; Binge; overconsumption of food; purging; purge
MeSH Terms: conditions — Bulimia Nervosa; Binge-Eating Disorder | interventions — Cognitive Behavioral Therapy; Exercise

STUDY DESIGN:
Intervention Model Description: Comparing treatment of cognitive behavioural therapy, with treatment of physical exercise and dietary therapy. All participants randomized to either of the two treatment offers. Waitlist serves as control group.
Who Masked: Outcomes Assessor
Masking Description: The one transferring results from lab's and questionaires to SPSS are blinded for group affiliation.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Behaviour Therapy (Experimental): Treatment with small groups following a modified protocol first described by Fairburn 2008
  Interventions: Behavioral: Cognitive Behaviour Therapy
- Physical activity and dietary therapy (Experimental): Treatment with guided physical activity and dietary therapy in small groups
  Interventions: Behavioral: Physical Activity and Dietary Therapy

INTERVENTIONS:
Behavioral: Cognitive Behaviour Therapy — Following group-modified protocol for cognitive behavioral therapy, CBT, first described by Fairburn 2008, modified by Modum Bad, Norway.
  Other Names: CBT-ED; CBT-enhanced; CBT-e
  Arms: Cognitive Behaviour Therapy
Behavioral: Physical Activity and Dietary Therapy — Guided physical activity and dietary therapy, to (re-)introduce a more healthy lifestyle and help stabilizing a healthy weight. A detailed manual will be published.
  Other Names: PADT; FAKT; PED-t
  Arms: Physical activity and dietary therapy

SUMMARY:
"Eating disorders" includes anorexia nervosa, bulimia nervosa, binge eating and other specified feeding or eating disorder (OSFED). Common to all is the intensively occupation to control food intake, body image and body weight. Most people with this kind of disorder don't reach for professional help, or there may be more than 4 years before they do. Cognitive behavior therapy is the foremost method of treatment of eating disorders, but up to 30-50% of the patients don't respond to this. The investigators find it important to identify science based alternatives of therapy, as this may reduce the health concern, and broaden the choice of therapy methods. A former study by Sundgot-Borgen et al in 2002, found guided physical activity to reduce symptoms of bulimia nervosa just as good as the traditional cognitive therapy.

The primary objective of the project is to see whether the combination of physical exercise and dietary therapy is more effective in treating eating disorders, than cognitive therapy.

Secondly, the investigators want to see whether there are any differences with regard to the individual satisfaction of treatment method, and to associated costs. Interviews with a sufficient number of participants from the PED-t arm to meet data saturation criteria, and all theraphists in the new treatment offer, will give uniqe insight to experiences with the treatment method and the delivery of treatment.

DETAILED DESCRIPTION:
Subjects are recruited through primary doctors, social media and newspapers, and will be included continuously by screening interviews. There will be a randomization into two treatment groups (cognitive behavior, or physical activity and nutrition education) to be followed for 16 weeks. Each week includes one meeting of group therapy (90 minutes) and homework related to treatment, and for 4 weeks midway there will be two therapy meetings pr week (a total of 20 meetings). Post tests are planned at week 17, and at 6, 12, and 24 months after treatment.

Participants reqruited during ongoing treatment groups are placed on a waitlist, serving as controls to the treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Women,
* BMI 17,5-35,
* Age of 18-40 years,
* DSM-5 criteria of bulimia nervosa,
* DSM-5 criteria of Binge eating disorder
* Living nearby Norwegian School of Sports Sciences, NSSS, in Oslo (Norway)

Exclusion Criteria:

* Age <18 and >40 years
* BMI <17,5 and >35
* Pregnancy
* Competing/experienced athlete
* Anorexia nervosa
* Currently, or during the past 2 years, in active treatment with cognitive therapy
* Other personality disturbances
* Suicidality

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Effectiveness of treatment, evaluated through the change in symptoms of eating disorder | Pre-test in week 0, Post-tests (week 17), and at 6, 12, and 24 months after intervention.
  Change in ED-symptoms are evaluated through screening and surveys: EDE-questionaire (Episodes of binge eating, episodes of purging, concern for body weight and appearance)(Fairburn, 2008), Clinical Impairment Assessment (CIA) (Fairburn, 2008), Eating Disorder Inventory-3 (EDI) (Garner, 2004), Eating Disturbance Scale (EDS-5) (Rosenvinge et al., 2000), DSM-5 (APA, 2013)

SECONDARY OUTCOMES:
Expectations of treatment method for eating disorders | Pre-test
  Interview on the expectations the patients have to the specified treatment method of eating disorders (arm of intervention) EPDEX (Clinton 2001)
Experiences of the treatment method for eating disorders | Post-test (week 17)
  Interview on the experiences the patients have to the specified treatment method of eating disorders (arm of intervention), EPDEX (Clinton 2001)
Associated cost with treatment method | Pre-test
  Calculation of the directly and indirectly cost related to treatment method
Associated cost with treatment method | Post-test (week 17)
  Calculation of the directly and indirectly cost related to treatment method
Associated cost With treatment method | Post-test (by 6th month post-treatment)
  Calculation of the directly and indirectly cost related to treatment method
Associated cost With treatment method | Post-test (by 12th month post-treatment)
  Calculation of the directly and indirectly cost related to treatment method
Associated cost with treatment method | Post-test (by 24th month post-treatment)
  Calculation of the directly and indirectly cost related to treatment method
Global measurement of general psychopathology | Pre-treatment
  Beck's Anxiety Inventory (BAI), Beck Depression Inventory (BDI), QoL (Diener), Utrecht Coping List, Resilience Scale for Adults, the outcome rating scale (ORS), the three-factor eating questionnaire (TFEQ), Binge eating Scale (BES), Cantril's Ladder, Exercise dependency test, compulsice exercise test
Global measurement of general psychopathology | Post-treatment (week 17)
  Beck's Anxiety Inventory (BAI), Beck Depression Inventory (BDI), QoL (Diener), Utrecht Coping List, Resilience Scale for Adults, the outcome rating scale (ORS), the three-factor eating questionnaire (TFEQ), Binge eating Scale (BES), Cantril's Ladder, Exercise dependency test, compulsice exercise test
Global measurement of general psychopathology | Post-treatment (by the 6th month post-treatment)
  Beck's Anxiety Inventory (BAI), Beck Depression Inventory (BDI), QoL (Diener), Utrecht Coping List, Resilience Scale for Adults, the outcome rating scale (ORS), the three-factor eating questionnaire (TFEQ), Binge eating Scale (BES), Cantril's Ladder, Exercise dependency test, compulsice exercise test
Global measurement of general psychopathology | Post-test (by 12th month post-treatment)
  Beck's Anxiety Inventory (BAI), Beck Depression Inventory (BDI), QoL (Diener), Utrecht Coping List, Resilience Scale for Adults, the outcome rating scale (ORS), the three-factor eating questionnaire (TFEQ), Binge eating Scale (BES), Cantril's Ladder, Exercise dependency test, compulsice exercise test
Global measurement of general psychopathology | Post-test (by 24th month post-treatment)
  Beck's Anxiety Inventory (BAI), Beck Depression Inventory (BDI), QoL (Diener), Utrecht Coping List, Resilience Scale for Adults, the outcome rating scale (ORS), the three-factor eating questionnaire (TFEQ), Binge eating Scale (BES), Cantril's Ladder, Exercise dependency test, compulsice exercise test
Group climate | week 1-16
  coerciveness scale from Therapeutic Factor Inventory (Lese & MacNair-Semands, 2000).
Working AIliance | week 1-16
  Working AIliance Inventory (Horwath & Greenberg, 1989)
Experiences of the treatment method for eating disorders | Post-test (6 months)
  Interview on the experiences the patients have to the specified treatment method of eating disorders (arm of intervention) (Clinton 2001)
Experiences of the treatment method for eating disorders | Post-test (by 12th month post-treatment)
  Interview on the experiences the patients have to the specified treatment method of eating disorders (arm of intervention) (Clinton 2001)
Experiences of the treatment method for eating disorders | Post-test (by 24th month post-treatment)
  Interview on the experiences the patients have to the specified treatment method of eating disorders (arm of intervention) (Clinton 2001)
Change in eating disorder behavior and cognitions related to body figure and bodyweight | Week 1-16 during treatment
  Evaluation after each therapy session on progress in reducing eating disordered behaviour (binging and purging) and on changes of cognitions on body figure and -weight

OTHER OUTCOMES:
Change in muscular strength | Pretest (week 0), post-test (week 17) and at 6, 12 and 24 months after treatment
  Status of 1 repetition maximum, 1RM, muscular strength in squats, bench press and seated row
Change in cardiovascular endurance | Pre-test in week 0, Post-tests ( week 17), and at 6, 12 and 24 months after intervention.
  CPET: with the use of modified Balke Treadmill performance evaluation test, The Borg scale (Borg, 1982)
Change in bone mineral density | Pre-test in week 0, Post-test (week 17) and 6, 12, and 24 months post-treatment
  DXA (Dual-energy X-ray absorptiometry)
Change in body weight and bodycomposition | Pre-test and post-test (week 17) and at 6,12,18 and 24 months post-treatment
  DXA (dual-energy x-ray absorptiometry) (weekly weight registration will also be kept in each arm of treatment)
Change in nutritional status | Pre-test, in week 8 of treatment, post-test (week 17) and at 6,12,18 and 24 months post-treatment
  Blood test to identify nutritional status of iron, folate, cholesterol and triglycerides, ApoA, ApoB and vitamin-D, folic acid
Change in hormonal status | Pre-test, week 8 of treatment, post-test (week 17) and at 6,12,18 and 24 months post-treatment
  Blood test to evaluate hormonal status of estradiol, progesterone, CTX, P1nP, insulin, leptin, TSH, T3, T4, FSH, LH, cortisol
Change in dietary and nutritional intake | Pre-test, each 3rd week in treatment (a total of 5 interviews), post-test (week 17), and post-treatment (6,12, and 24 months post-treatment)
  24 hour recall interview: interview on the intake of food and beverage during the past 24 hours.
Change in physical activity level | Pre-test in week 0, Post-test (week 17) and 6, 12, and 24 months post-treatment
  Wearing a GT3X-BT actigraph accelerometer for 7 consecutive days and making notes on daily activity in 30 minutes intervals
Interview: measure and explore patients experienced treatment satisfaction and outcome/benefits with PED-t. | Post treatment
  Qualitative approaches, such as in-depth interviews, will give additional insights into ED-patients' perspectives, notably experiences and satisfaction with the treatment. A sufficient number of participants to meet data saturation criteria are qualitatively interviewed.
  Data are analyzed in four steps within the framework of systematic text condensation (Malterud 2012).
Interview: What are the theraphists experiences of their contribution to the PED-t program | Post treatment
  Qualitative approaches, such as in-depth interviews, will give additional insights into the therapists' perspectives and experiences on delivering a new treatment offer for eating disorder.
  Data are analyzed in four steps within the framework of systematic text condensation (Malterud 2012).
Interview: What are the experiences of the participants who drop out of the PED-t program? | Post treatment
  Data are analyzed in four steps within the framework of systematic text condensation (Malterud 2012).

CONTACTS AND LOCATIONS:
Overall Officials: Jorunn Sundgot-Borgen, Professor, Study Chair — Norwegian School of Sports Sciences; Therese F Mathisen, PhDcandidate, Principal Investigator — Norwegian School of Sports Sciences; Jan Rosenvinge, Professor, Study Director — University of Tromso
Locations (1):
- Norwegian School of Sports Sciences, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sundgot-Borgen J, Rosenvinge JH, Bahr R, Schneider LS. The effect of exercise, cognitive therapy, and nutritional counseling in treating bulimia nervosa. Med Sci Sports Exerc. 2002 Feb;34(2):190-5. doi: 10.1097/00005768-200202000-00002. PMID 11828224
- [Derived] Mathisen TF, Sundgot-Borgen J, Rosenvinge JH, Bratland-Sanda S, Svendsen M, Pettersen G, Vrabel K, Friborg O. Metabolic profile in women with bulimia nervosa or binge-eating disorder before and after treatment: secondary analysis from the randomized PED-t trial. Eat Weight Disord. 2023 Apr 27;28(1):41. doi: 10.1007/s40519-023-01567-y. PMID 37103592
- [Derived] Mathisen TF, Rosenvinge JH, Friborg O, Vrabel K, Bratland-Sanda S, Pettersen G, Sundgot-Borgen J. Is physical exercise and dietary therapy a feasible alternative to cognitive behavior therapy in treatment of eating disorders? A randomized controlled trial of two group therapies. Int J Eat Disord. 2020 Apr;53(4):574-585. doi: 10.1002/eat.23228. Epub 2020 Jan 16. PMID 31944339
- [Derived] Pettersen G, Rosenvinge JH, Skomakerstuen T, Sordal S, Mathisen TF, Sundgot-Borgen J. Patient expectations of a new treatment for eating disorders combining guided physical exercise and dietary therapy: an interview study of women participating in a randomised controlled trial at the Norwegian School of Sport Sciences. BMJ Open. 2019 Apr 20;9(4):e025344. doi: 10.1136/bmjopen-2018-025344. PMID 31005919
- [Derived] Mathisen TF, Bratland-Sanda S, Rosenvinge JH, Friborg O, Pettersen G, Vrabel KA, Sundgot-Borgen J. Treatment effects on compulsive exercise and physical activity in eating disorders. J Eat Disord. 2018 Dec 13;6:43. doi: 10.1186/s40337-018-0215-1. eCollection 2018. PMID 30559966
- [Derived] Mathisen TF, Rosenvinge JH, Friborg O, Pettersen G, Stensrud T, Hansen BH, Underhaug KE, Teinung E, Vrabel K, Svendsen M, Bratland-Sanda S, Sundgot-Borgen J. Body composition and physical fitness in women with bulimia nervosa or binge-eating disorder. Int J Eat Disord. 2018 Apr;51(4):331-342. doi: 10.1002/eat.22841. Epub 2018 Feb 23. PMID 29473191
- [Derived] Mathisen TF, Engen KM, Sundgot-Borgen J, Stensrud T. Evaluation of a short protocol for indirect calorimetry in females with eating disorders and healthy controls. Clin Nutr ESPEN. 2017 Dec;22:28-35. doi: 10.1016/j.clnesp.2017.09.003. Epub 2017 Oct 5. PMID 29415831
- [Derived] Bakland M, Sundgot-Borgen J, Wynn R, Rosenvinge JH, Stornaes AV, Pettersen G. Therapists' experiences with a new treatment combining physical exercise and dietary therapy (the PED-t) for eating disorders: an interview study in a randomised controlled trial at the Norwegian School of Sport Sciences. BMJ Open. 2018 Jan 11;8(1):e019386. doi: 10.1136/bmjopen-2017-019386. PMID 29330176
- [Derived] Pettersen G, Rosenvinge JH, Bakland M, Wynn R, Mathisen TF, Sundgot-Borgen J. Patients' and therapists' experiences with a new treatment programme for eating disorders that combines physical exercise and dietary therapy: the PED-t trial. A qualitative study protocol. BMJ Open. 2018 Jan 8;8(1):e018708. doi: 10.1136/bmjopen-2017-018708. PMID 29317417
- [Derived] Pettersen G, Sordal S, Rosenvinge JH, Skomakerstuen T, Mathisen TF, Sundgot-Borgen J. How do women with eating disorders experience a new treatment combining guided physical exercise and dietary therapy? An interview study of women participating in a randomised controlled trial at the Norwegian School of Sport Sciences. BMJ Open. 2017 Dec 19;7(12):e018588. doi: 10.1136/bmjopen-2017-018588. PMID 29259061
- [Derived] Mathisen TF, Rosenvinge JH, Pettersen G, Friborg O, Vrabel K, Bratland-Sanda S, Svendsen M, Stensrud T, Bakland M, Wynn R, Sundgot-Borgen J. The PED-t trial protocol: The effect of physical exercise -and dietary therapy compared with cognitive behavior therapy in treatment of bulimia nervosa and binge eating disorder. BMC Psychiatry. 2017 May 12;17(1):180. doi: 10.1186/s12888-017-1312-4. PMID 28494809
- See also: Norwegian School of Sports Sciences — http://www.nih.no/en/
- See also: The Norwegian Women's Public Health Association — http://www.sanitetskvinnene.no/
- See also: University of Tromsø — http://en.uit.no/startsida
- See also: Modum Bad — http://translate.google.com/translate?hl=no&langpair=no%7Cen&u=http://www.modum-bad.no/
- See also: Recruitment webpage — http://nihfakt.blogspot.no/